CLINICAL TRIAL: NCT04616963
Title: F/TAF Switch Study for Transgender Individuals for HIV Pre-exposure Prophylaxis (TAF4TRANS)
Brief Title: Emtricitabine/Tenofovir Alafenamide Switch Study for Transgender Individuals for HIV Pre-exposure Prophylaxis
Acronym: TAF4TRANS
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: CCTG 605
Record Dates: First submitted 2020-07-13; First posted 2020-11-05 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hiv; Hormone Therapy
Keywords: Pre-exposure Prophylaxis; PrEP; Hormone Therapy; HT
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Intervention Model Description: Following Phase I lead-in, all participants will continue PrEP with fixed dose combination daily oral F/TAF substituting for F/TDF in Phase II. Participants will continue to receive PrEP in accordance with standardized comprehensive methods of prescribing, which includes risk reduction counseling, adherence counseling, and clinical assessments with safety monitoring, as well as HIV and STI screening. Participants will receive daily adherence-supporting text message reminders through 12 weeks after F/TAF initiation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FTC 200 mg / TDF 300 mg and FTC 200 mg / TAF 25 mg (Other): Phase I: Participants will continue or initiate F/TDF for PrEP for a minimum 12-week lead-in period prior to switching to F/TAF.
  Phase II: Participants will be switched to study-provided F/TAF for PrEP until 48 weeks after initiation. Participants will receive study treatment for the duration of the study unless they meet criteria for discontinuation.
  Interventions: Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet 200/300 mg; Drug: Emtricitabine Tenofovir Alafenamide 200/25 mg

INTERVENTIONS:
Drug: Emtricitabine / Tenofovir Disoproxil Oral Tablet 200/300 mg — Following Phase I lead-in, all participants will continue PrEP with fixed dose combination daily oral F/TAF substituting for F/TDF in Phase II. Participants will continue to receive PrEP in accordance with standardized comprehensive methods of prescribing, which includes risk reduction counseling, adherence counseling, and clinical assessments with safety monitoring, as well as HIV and STI screening. Participants will receive daily adherence-supporting text message reminders through 12 weeks after F/TAF initiation.
  Other Names: Truvada 200Mg-300Mg Tablet
Drug: Emtricitabine Tenofovir Alafenamide 200/25 mg — Following Phase I lead-in, all participants will continue PrEP with fixed dose combination daily oral F/TAF substituting for F/TDF in Phase II. Participants will continue to receive PrEP in accordance with standardized comprehensive methods of prescribing, which includes risk reduction counseling, adherence counseling, and clinical assessments with safety monitoring, as well as HIV and STI screening. Participants will receive daily adherence-supporting text message reminders through 12 weeks after F/TAF initiation
  Other Names: Descovy 200Mg-25Mg Tablet

SUMMARY:
The purpose of this study is to evaluate Pre-Exposure Prophylaxis (PrEP) levels in transgender-identifying or gender non-binary individuals taking versus not taking gender affirming hormone therapy. Subjects who have previously taken F/TDF as PrEP will continue with a fixed dose combination of daily oral F/TAF substituting for F/TDF. Subjects will receive the iTAB text messaging adherence reminders to provide personalized, automated text messages to support and monitor adherence that will vary by participant choice until 12 weeks after switching medication. This study will enroll 60 individuals to take F/TAF as PrEP for 48 weeks.

DETAILED DESCRIPTION:
This is a two-phased prospective switch study of 60 transgender individuals who are eligible for Truvada® (Emtricitabine/Tenofovir Disoproxil Fumarate) F/TDF PrEP and who are willing to switch to Descovy® (Emtricitabine/Tenofovir Alafenamide) F/TAF for 48 weeks. The purpose of the current study is to contribute safety and efficacy data to support the use of F/TAF in transgender/non-binary individuals. The current study leverages existing studies in trans/non-binary populations (e.g. CCTG 603; HRPP#161807) funded by the California HIV/AIDS Research Program (CHRP).

The dosage for Phase I is FTC 200 mg / TDF 300 mg. The dosage for Phase II is FTC 200 mg / TAF 25 mg. TDF/FTC is FDA approved for use as PrEP in adults and adolescents at risk for HIV-1. F/TAF has received approval by the FDA for use as PrEP as of October 3rd, 2019 except for those having receptive vaginal sex. The FDA has yet to approve F/TAF for use in those having receptive vaginal sex due to a lack of clinical research studies specific to the population. Participants will be advised that if they decide to have receptive vaginal sex while taking F/TAF, they should use another method of protection such as condoms.Eligibility criteria will be based on the CDC guidance for PrEP use in transgender persons. All participants must be confirmed HIV-negative (either by rapid test or Ag/Ab test), must have acceptable safety laboratory values, and must currently be taking or will initiate F/TDF by the Screening/Baseline visit. Participants will have a 12-week lead-in period prior to switching to F/TAF. At the Switch Visit, participants will be instructed to substitute F/TDF with F/TAF for PrEP for 48 weeks. Regular follow-up evaluations will occur at Weeks 12, 24, 36, and 48.

Participants will receive health education, clinical assessments, laboratory safety monitoring, STI and HIV screening, standard HIV risk reduction and adherence counseling, assessment of psychosocial barriers, and completion of a computer-based self-report survey that includes assessments of adherence and risk behaviors. Intracellular TFV-DP quantification will be performed in retrospect on batched, banked samples and additional banked specimens will be frozen for future use. Adherence by TFV-DP concentrations and self-reported measures will be used for the primary and secondary analyses of the study. Additional outcomes for the study will include changes in risk behavior and determinants of PrEP adherence.

This study will continue iTAB, a daily text message support system for adherence up until 12 weeks after F/TAF switch. As needed, the study will provide a) subject reimbursement to pay for unlimited text messaging and/or b) an appropriate cell phone if a subject does not have one. Daily dosing text message reminders will be sent for the duration of the study. Both reminder timing and content can be individualized. Participants have selected 15 personal reminders from a list of pre-determined reminders that cover various themes shown to be effective in improving adherence (e.g., social support, loss frame, health gain, etc.) as developed through focus groups and targeted group feedback. These messages can be modified and the patient can choose to create their own reminders if they prefer. These reminder times can vary for different days of the week to accommodate for changes in schedule (e.g., 8 M-F, and 10 AM on Sat/Sun). Once the time is identified, the text reminder system is automated. Patients will confirm medication taking via text responses to the personalized reminders.

ELIGIBILITY:
Inclusion Criteria:

1. Transgender or non-binary, defined as identifying with a gender differently from sex assigned at birth
2. Age 18 years or older
3. Currently eligible to take F/TDF for PrEP and willing to switch to F/TAF
4. Negative for HIV infection
5. Acceptable renal function as measured by calculated creatinine clearance of at least 60 mL/min by the Cockcroft-Gault formula in the past 30 days

Exclusion Criteria:

1. Unable to give informed consent
2. Active hepatitis B defined by a positive hepatitis B surface antigen (HBsAg)
3. Substantial medical condition that, in the opinion of the investigator, would preclude participation, as defined by

   * gastrointestinal condition that would impair absorption of study drugs
   * known condition of reduced bone density (e.g. osteoporosis or osteogenesis imperfect) that significantly elevate the risk of bone fracture
   * neurological or severe psychiatric condition that would significantly impair the ability to adhere to PrEP
   * tubular or glomerular kidney disease that could be exacerbated by tenofovir
   * other medical condition that would unacceptably increase the risk of harm from study drug or significantly impair the ability to adhere to PrEP
4. Suspected sensitivity or allergy to the study drug or any of its components
5. Currently using an essential product or medication that interacts with the study drug such as the following:

   * other antiretroviral agent other than F/TDF (including nucleoside analogs, non-nucleoside reverse transcriptase inhibitors, integrase inhibitors, protease inhibitors or investigational antiretroviral agents)
   * agents with known nephrotoxic potential:

     * aminoglycoside antibiotics (including gentamicin)
     * IV amphotericin B
     * cidofovir
     * cisplatin
     * foscarnet
     * IV pentamidine
     * IV vancomycin
     * oral or IV gancyclovir
     * other agents with significant nephrotoxic potential

       - drugs that slow renal excretion
     * probenecid

       - immune system modulators
     * systemic chemotherapeutic agents (i.e. cancer treatment medications)
     * ongoing systemic corticosteroids (with the exception of short courses of tapering steroid doses for asthma or other self- limited condition).
     * interleukin-2 (IL-2)
     * interferon (alpha, beta, or gamma)

       - other agent known to have a significant interaction with TDF, TAF, or FTC
     * the following table includes medications/herbal supplements to be excluded or should be used with caution while participants are taking study drugs due to potential drug-drug interactions with F/TAF.
6. Proteinuria 2+ or greater by urine dipstick
7. Pregnancy (if applicable)
8. Other condition that, in the opinion of the investigator, would put the participant at risk, complicate interpretation of study outcome data, or would otherwise interfere with participation or achieving the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Measuring tenofovir diphosphate (TFV-DP) concentrations | Baseline-48 weeks
  Analysis will be performed on the primary outcome of TFV-DP levels by HT status. Comparison of those on and off HT will be done be t-test. Additional sub-analysis of the primary will stratify by HT type and using both concentrations of TFV-DP and estradiol levels test for correlation. Also cut offs for adherence consistent with 4 doses a week and 7 doses a week will be compared between strata.

SECONDARY OUTCOMES:
Evaluating safety of F/TAF in transgender individuals compared to F/TDF: adverse events | Baseline-48 weeks
  Safety data will be reported for all participants during use of study drug and immediately after (30 days) completion (as treated analysis). Tables will summarize the number of serious adverse events, adverse events (Grade 1 or higher) over 48 weeks, and PrEP discontinuation due to adverse events.
Evaluating tolerability of F/TAF in transgender individuals compared to F/TDF. | Baseline-48 weeks
  Tolerability will be assessed using Likert scales for those that found favorable tolerability and greater between week 12 F/TDF and week 12 F/TAF.
  The Likert scale uses answers on a range of:
  * Strongly agree (maximum)
  * Agree
  * Neutral
  * Disagree
  * Strongly Disagree (minimum)
  A higher score (strongly agree) would indicate a better outcome for Descovy compared to Truvada.
Adherence to F/TAF in transgender individuals compared to F/TDF | Baseline-48 weeks
  Adherence will be assessed by comparing TFV-DP concentrations commensurate with i) 7 doses/week and ii) 4 doses/week; iii) TFV-DP levels as a continuous measure; and iv) self-reported adherence by text message over 48 weeks between participants on F/TDF versus participants on F/TAF
Evaluating serum creatinine between F/TDF and F/TAF. | Week 12
  Serum creatinine concentrations will be compared between Week 12 of F/TDF and Week 12 on F/TAF.
Evaluating calculated creatinine clearance between F/TDF and F/TAF. | Week 12
  Calculated creatinine clearance will be compared between Week 12 of F/TDF and Week 12 on F/TAF.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Morris, MD, Principal Investigator — UC San Diego AntiViral Research Center (AVRC)
Locations (1):
- UC San Diego AntiViral Research Center (AVRC), San Diego, California, United States

REFERENCES:
- [Derived] Patel N, Awdishu L, Burke LB, Vaingankar S, Chow K, Pacheco D, Silva J, Higgins N, Muttera L, Blumenthal J, Morris S. Comparison of Existing and New Race- and Sex-Free Kidney Function Equations in Transgender Adults without CKD. Clin J Am Soc Nephrol. 2025 Jul 22;20(9):1280-1282. doi: 10.2215/CJN.0000000688. No abstract available. PMID 40694414

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT04616963/Prot_SAP_000.pdf